CLINICAL TRIAL: NCT03559673
Title: Compassionate Use Program With Lacosamide in Patients With Partial-onset or Generalized Tonic-clonic Seizures ≥16 Years of Age Coming From the SP0994 Study
Brief Title: Compassionate Use Program With Lacosamide in Patients With Partial-onset or Generalized Tonic-clonic Seizures
Status: No longer available | Type: Expanded Access
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: EP0072
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Lacosamide

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Lacosamide — Patients will start on the individual Lacosamide (LCM) dose that they had reached at the completion of the previous monotherapy study. LCM will be administered orally twice daily in 2 divided doses.
  Other Names: Vimpat

SUMMARY:
The objective of this Compassionate Use Program (CUP) is to provide continued access to Lacosamide (LCM) for monotherapy use for patients who were receiving LCM in SP0993 and SP0994 at the time of study unblinding and close of SP0994, and who benefited from the treatment per investigator assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has completed the Termination Visit of SP0994 and has been treated with Lacosamide (LCM) monotherapy
* Patient is expected to benefit from participation in the Compassionate Use Program (CUP) with LCM monotherapy, in the opinion of the treating physician
* Patient is willing and able to comply with all program requirements
* Patient is informed of the details of this CUP, is given ample time and opportunity to ask questions and consider his/her participation in this CUP, and the patient or the legally authorized representative (LAR) has provided verbal consent to participate, and, if applicable to local regulations, has given written informed consent

Exclusion Criteria:

* Patient is receiving any investigational drugs or using any experimental devices in addition to LCM
* For countries where LCM is reimbursed: Patient requires another anti-epileptic drug (AED) for the treatment of seizures For countries where LCM is not reimbursed (or conditionally reimbursed: Belgium, Australia e.g.): Patient requires another AED for the treatment of seizures and qualifies for commercial LCM (and LCM is being reimbursed)
* Patient experienced emergence of a seizure type other than partial-onset or generalized tonic-clonic seizures, or occurrence of status epilepticus
* Patient developed second- or third-degree atrioventricular (AV) block or another clinically relevant change in medical condition (or electrocardiogram (ECG) or laboratory parameter)
* Patient having liver function test (LFT) results of transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) ≥3×ULN to <5×upper limit of normal (ULN)
* Patient has actual suicidal ideation or behavior
* Patient is experiencing an ongoing serious adverse event (SAE) and there is no expected benefit for him/her to continue on LCM treatment
* Female patient who is pregnant or nursing, and/or a woman of childbearing potential who is not surgically sterile, 2 year postmenopausal or does not practice one highly effective method of contraception (according to ICH guidance defined as those that result in a failure rate of less than 1 % per year when used consistently and correctly), unless sexually abstinent, for the duration of the study
* Patient was treated with carbamazepine controlled release (CBZ-CR) in SP0994

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)